CLINICAL TRIAL: NCT05640271
Title: Low-Dose Tocilizumab for Acute Chest Syndrome in Sickle Cell Disease
Brief Title: Tocilizumab for Acute Chest Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB22-0277
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease; Acute Chest Syndrome
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Chest Syndrome | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: All participants will receive tocilizumab 80 mg on one day and placebo (normal saline 50 mL) on another day, separated by 48 hours, and the order of these two doses will be randomized. Half the patients will receive tocilizumab at the time of acute chest syndrome diagnosis and subsequent randomization, and then that half will receive placebo two days later. The other half will receive placebo first and then tocilizumab two days later.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study statistician will generate randomizations using the method of permuted block randomization. The pharmacy will access the prepared randomization list via REDCap (a module separate from the clinical REDCap database) to guide tocilizumab versus placebo administration at the time of placing an inpatient order. Prior to randomization, the SpO2 to FiO2 ratio will be determined over an 8-hour period to serve as a baseline measure. Thus, randomization will be done at the time of placing the initial order for inpatient tocilizumab versus placebo, not at the time of enrollment. Patients, study investigators, and inpatient clinicians will all be blinded to the patient's randomized group assignment. Only the investigational pharmacy will be aware of the randomization arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Early Tocilizumab (Experimental): This arm will receive tocilizumab 80 mg at the time of acute chest syndrome diagnosis and subsequent randomization. Then, two days later, they will receive 50 mL of normal saline.
  Interventions: Drug: Tocilizumab
- Delayed Tocilizumab (Active Comparator): This arm will receive 50 mL of normal saline at the time of acute chest syndrome diagnosis and subsequent randomization. Then, two days later, they will receive tocilizumab 80 mg. Thus, this delayed arm will serve as a placebo comparator for the first 48 hours and then as an active comparator for the remaining duration on study.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 80 mg IV dose (one time per patient)

SUMMARY:
The investigators are evaluating the role of a low dose of tocilizumab in treating acute chest syndrome in patients with sickle cell disease. Tocilizumab inhibits interleukin-6 (IL-6) receptors and is used to treat rheumatoid arthritis and severe cytokine release syndrome, which can be seen with chimeric antigen receptor T-cell (CAR-T) therapy, and it is also authorized for treatment of COVID-19. Since IL-6 levels are elevated in the sputum of patients with acute chest syndrome, the investigators are hopeful that this will be an effective strategy. The investigators will be looking at how a low dose of tocilizumab affects oxygen status, clinical outcomes, and laboratory markers in patients admitted to the hospital with acute chest syndrome.

DETAILED DESCRIPTION:
In this randomized, placebo-controlled, double-blinded phase II study, enrolled patients admitted to the University of Chicago who are diagnosed with acute chest syndrome will receive one dose of tocilizumab 80 mg IV and one normal saline placebo dose. The order of these doses will be randomized at a 1:1 ratio. After collecting oxygenation data as a baseline for 8 hours, patients will then receive tocilizumab versus placebo as their early dose and then the opposite (placebo versus tocilizumab) 48 hours later. Clinical, laboratory, and patient-reported outcome data will be collected during their admission and compared between arms.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 12 years of age
* Prior diagnosis of sickle cell disease (Hb SS, Hb SC, Hb Sb+, and Hb Sb0)

Exclusion Criteria:

* Pregnant patients or breastfeeding mothers.
* Prior treatment with gene therapy or a stem cell transplant.
* Current enrollment in a clinical trial involving an FDA-regulated drug or biologic.
* Current neutropenia (absolute neutrophil count < 1000/mm^3)
* Current thrombocytopenia (platelet count < 50,000 mm^3)
* Aspartate aminotransferase (AST) or alanine transaminase (ALT) > 10 times the upper limit of normal (ULN)
* History of tuberculosis (TB).
* Positive purified protein derivative (PPD) TB screening test.
* On active therapy with a Bruton's tyrosine kinase-targeted agent, which include the following: Acalabrutinib, Ibrutinib, Zanubrutinib
* On active therapy with a JAK2-targeted agent, which include the following: Baricitinib, Ruxolitinib, Tofacitinib, Upadacitinib
* Any of the following biologic immunosuppressive agent (and any biosimilar versions thereof) administered in the past 6 months:

Abatacept, Adalimumab, Alemtuzumab, Atezolizumab, Belimumab, Blinatumomab, Brentuximab, Certolizumab, Daratumumab, Durvalumab, Eculizumab, Elotuzumab, Etanercept, Gemtuzumab, Golimumab, Ibritumomab, Infliximab, Inotuzumab, Ipilimumab, Ixekizumab, Moxetumomab, Nivolumab, Obinutuzumab, Ocrelizumab, Ofatumumab, Pembrolizumab, Polatuzumab, Rituximab, Sarilumab, Secukinumab, Tocilizumab, Tositumumab, Tremelimumab, Urelumab, Ustekinumab

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Time-weighted SaO2/FiO2 ratio | Total of 4 days (Day 0 to Day 4)
  Oxygenation data will be obtained as part of routine clinical care. All changes in pulse oximetry measurement that are documented in the chart will be recorded in an oxygen saturation case report form with the date and time from Day 0 to Day 4. These peripheral oxygen saturation (SpO2) measurements will serve as surrogates for SaO2. Additionally, all changes in the route of supplemental oxygen delivery, rate of supplemental oxygen delivery, and fraction of inspired oxygen (FiO2) will be recorded in a corresponding case report form with the date and time from Day 0 to Day 4. The time-weighted SaO2/FiO2 ratio, our primary endpoint, will be calculated based on these two case report forms.

SECONDARY OUTCOMES:
Red cell exchange transfusion rate | Total of 9 days (Day 0 to Day 8)
  As part of routine clinical care by the inpatient team, patients may receive a red cell exchange transfusion. The study team will assess if participants received any exchange transfusions from Day 0 to Day 8, and if so, they will record the date of the first exchange transfusion and the total number of units transfused during that time period.
Intensive Care Unit (ICU) transfer rate | Total of 9 days (Day 0 to Day 8)
  Patients will be assessed for if they were admitted directly to the intensive care unit (ICU) or if they were transferred from the general medicine floor to the ICU between Day 0 and Day 8. The date of transfer to the ICU will be recorded if applicable.
Length of stay | Up to 3 months (Admission Date to Discharge Date)
  Patients will be assessed for their admission and discharge dates. Length of stay will be calculated based on those two dates.
Readmission rate | Total of 29 days (Discharge Date to 28 days after discharge)
  Patients will be assessed for readmission for 28 days from discharge. Readmission will be assessed at the University of Chicago as well as through any linked hospitals through Care Everywhere within the electronic medical record system. The date of readmission will be recorded if applicable.
Mortality rate | Total of 29 days (Day 0 to Day 28)
  Patients will be assessed for mortality from Day 0 to Day 28. The date of death will be recorded if applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Austin Wesevich, MD, Study Director — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No